CLINICAL TRIAL: NCT01870557
Title: Markers of Bone Status in Diabetes Mellitus (Type 1 and Type 2)
Acronym: Diabone
Status: Completed | Type: Observational
Sponsor: Jakob Starup Linde (Other)
Responsible Party: Sponsor-Investigator, Jakob Starup Linde, MD, Aarhus University Hospital
Organization: University of Aarhus (Other)
Other Study IDs: 36777
Record Dates: First submitted 2013-05-29; First posted 2013-06-06 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Diabetes Mellitus; Osteoporosis; Osteopenia
Keywords: Diabetes Mellitus; Bone; Bone Status; Glycemic Markers; Osteoporosis; Osteopenia
MeSH Terms: conditions — Diabetes Mellitus; Osteoporosis; Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum Plasma EDTA Plasma Heparin Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Diabetes Mellitus type 1: n=100
- Diabetes Mellitus type 2: n=100

SUMMARY:
Objective To collate the bone status in type 1 and type 2 diabetics using biochemical markers and bone scans.

Methods:

This is a multicenter trial involving the University Hospitals of three major danish cities: Aalborg, Aarhus and Odense. The trial is of cross-sectional design and consists of examinations including:

* Blood samples to analyze bone markers, glycemic state, kidney function and sex-hormones.
* 24 hour urine sample to analyze bone markers and kidney function.
* Bone scans including dual energy x-ray absorptiometry (DXA) and high resolution peripheral quantitative computed tomography (HRpQCT) to evaluate Bone Mineral Density, t-score and bone structure.

Participants:

100 type 1 diabetics and 100 type 2 diabetics recruited from outpatient clinics at Aalborg, Aarhus and Odense, general practitioners and flyers.

DETAILED DESCRIPTION:
Diabetes Mellitus and Osteoporosis are common conditions. Patients with Diabetes Mellitus are known to have more fractures than their non-diabetic counterparts. However bone mineral density (BMD) which is the most commonly used measure of fracture risk seems to be insensitive in diabetes, thus BMD is lowered in type 1 diabetes but not enough to explain an almost seven fold in fracture risk. BMD is increased in type 2 diabetes although they still have an increased fracture risk.

The investigators investigate this paradox in diabetes by assessing type 1 and type 2 diabetes patients bone status by blood- and urine samples (assessing markers of bone- and glycemic state) and two types of bone scans comprising of DXA and HRpQCT scan.

The diabetes mellitus patients are recruited from outpatients clinics in the three study sites (Aalborg, Aarhus and Odense) as well as general practitioners and by flyers and adds.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or type 2 diabetes.
* Age ≥ 50 years.
* Unaltered treatment of diabetes during the previous six months (no changes in drugs, but an increase or decrease in dose is accepted) and HbA1c is stable with a level of ± 1 in the same period.
* HbA1c level≥ 7 % through the previous six months.
* BMI between 19 og 35.

Specific inclusion criteria for type 2 diabetes:

* Either treatment with metformin, sulfonylureas, dipeptidyl peptidase IV (DPP IV) inhibitors or glucagon-like peptide 1 (GLP-1) analogs.
* Treatment with insulin and insulin in the combination with metformin, sulfonylureas, DPP IV inhibitors or GLP-1 analogs.

Exclusion Criteria:

* HbA1C > 10%
* Pregnancy.
* Metal implanted at both ankles and wrists.
* Patients treated with: Antiresorptive (incl. hormone replacement therapy) or bone anabolic treatment, glucocorticoids, lithium and anticonvulsives.
* Patients with a bone disease other than osteoporosis.
* Vertebral fracture visible by vertebral fracture assessment (VFA).
* Patients with renal disease defined by estimated glomerular filtration rate(eGFR) < 50.
* Other medical disease in unstable phase (fx. cancer, hyperthyroidism).
* Heart failure; New York Heart Association (NYHA) class IV.
* Patients which the investigator does not believe is fit to participate in the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 Diabetes Mellitus patients. 100 with type 1 diabetes and 100 with type 2 diabetes. Of the 100 type 2 diabetes patients half should be treated with insulin (n=50) and the other half treated with other oral antidiabetics and not insulin.
Sampling Method: Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
HbA1c | Baseline
  Long term blood glucose evaluation
Bone Mineral Density (t-score) | Baseline

SECONDARY OUTCOMES:
Biochemical Bone Markers | Baseline
Sex-hormones | Baseline
Electrolytes | Baseline
Vitamin D (25ODH /1,25OHD) | Baseline
Results from the HRpQCT scan including Trabecular and Cortical state | Baseline
  Not available for participants at center Aalborg
Markers of fat tissue and glycemic status | Baseline
  Including Insulin level, adiponectin
Verterbral fracture assessment | Baseline
  A part of the DXA if vertebral fracture assessment is available. For patients at center Aalborg this will be evaluated through X-ray.
Lifestyle and Medical history | Baseline
  Assessed by structured interview and questionnaire. Information on alcohol consumption, smoking, pharmaceutical use, diabetes complications, diabetes duration, physical activity, previous fractures are collected.

OTHER OUTCOMES:
urine creatinine albumin ratio | Baseline
  Collected by both 24 hour urine samples and a urine sample.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Vestergaard, Professor MD PhD DrMedSc, Principal Investigator — Aalborg University Hospital; Kim Brixen, Professor MD PhD DrMedSc, Principal Investigator — Odense University Hospital; Søren Gregersen, MD PhD, Study Chair — Aarhus University Hospital; Bente Lomholt Langdahl, Professor MD PhD DrMedSc, Study Chair — Aarhus University Hospital; Ellen-Magrethe Hauge, MD PhD, Study Chair — Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Department of Endocrinology, Aalborg University Hospital, Aalborg
  - Department of Endocrinology and Internal Medicine, Aarhus University Hospital, Aarhus

REFERENCES:
- [Derived] Starup-Linde JK, Viggers R, Langdahl B, Gregersen S, Lykkeboe S, Handberg A, Vestergaard P. Associations of Circulating Osteoglycin With Bone Parameters and Metabolic Markers in Patients With Diabetes. Front Endocrinol (Lausanne). 2021 Mar 15;12:649718. doi: 10.3389/fendo.2021.649718. eCollection 2021. PMID 33790870
- [Derived] Starup-Linde J, Lykkeboe S, Gregersen S, Hauge EM, Langdahl BL, Handberg A, Vestergaard P. Bone Structure and Predictors of Fracture in Type 1 and Type 2 Diabetes. J Clin Endocrinol Metab. 2016 Mar;101(3):928-36. doi: 10.1210/jc.2015-3882. Epub 2016 Jan 12. PMID 26756117
- [Derived] Starup-Linde J, Lykkeboe S, Gregersen S, Hauge EM, Langdahl BL, Handberg A, Vestergaard P. Differences in biochemical bone markers by diabetes type and the impact of glucose. Bone. 2016 Feb;83:149-155. doi: 10.1016/j.bone.2015.11.004. Epub 2015 Nov 10. PMID 26555635